CLINICAL TRIAL: NCT06670716
Title: VERY BRIEF SPEECH and MEMORY ASSESSMENTS USING ALBA a PICNIR TESTS and DELIRIUM ASSESSMENTS USING CAM-ICU and ICDSC TESTS in PATIENTS SHORTLY AFTER the STROKE
Brief Title: BRIEF COGNITIVE and DELIRIUM ASSESSMENTS in STROKE PATIENTS
Acronym: COGISTROKE
Status: Active, not recruiting | Type: Observational
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Magda Michalovová, Medical doctor, Faculty Hospital Kralovske Vinohrady
Other Study IDs: EK-VP l05l00l2024
Record Dates: First submitted 2024-07-29; First posted 2024-11-01 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-07

CONDITIONS: Stroke Acute
Keywords: stroke; kognitive function; delirium
MeSH Terms: conditions — Stroke; Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with schemic or hemorrhagic CVA: Patients admitted to the monitored bed of the neurological ICU for ischemic or hemorrhagic CVA, with the possibility of an initial examination within 24 hours of admission (not the onset of CVA), and with an anticipated length of hospitalization longer than five days, will be included in the study.
  Interventions: Other: Examination by a speech therapist; Diagnostic Test: Cognitive examination; Other: Examination of delirium; Other: History taking

INTERVENTIONS:
Other: Examination by a speech therapist — MASTcz test
Diagnostic Test: Cognitive examination — ALBA test, PICNIR test
Other: Examination of delirium — CAM-ICU and ICDSC questionnaire
Other: History taking — The first page includes several sections: personal information, pre-stroke history, time-related data, neurological deficit data, radiological evaluation, pre-admission and admission treatment, and a medical examination focused on motor and speech impairments. The third page will document the physician's delirium examination and the speech therapy assessment. A questionnaire will be given to the relatives or close persons of the patients to fill out in order to collect systematic personal and pre-stroke anamnestic data and to assess the presence of dementia signs before the stroke using the Blessed Dementia Scale (BDS) questionnaire. All pages of the record form and the Questionnaire for Relatives are included in the appendices.

SUMMARY:
The aim of the project is to validate the ALBA and PICNIR tests for the easy detection of memory and speech disorders in patients after a stroke. Patients, after their first stroke, with the possibility of initial clinical evaluation within 24 hours of admission to the Neurology Clinic ICU, will undergo a neurological examination, cognitive tests using the ALBA and PICNIR tests, delirium tests using the CAM-ICU and ICDSC tools, and a speech therapy test using the MASTcz tool. If possible, these will be conducted simultaneously in one half-day. A similar structured examination will take place within five days, with a tolerance of one day. Upon demonstrating utility, doctors will be able to utilize the very brief ALBA and POBAV methods for detecting memory and speech disorders in post-stroke patients in clinical practice.

DETAILED DESCRIPTION:
Speech and motor production disorders are easily recognizable or examinable symptoms of stroke (Cerebrovascular Accident - CVA). In contrast, memory disorders are rarely examined, primarily within research studies rather than routine clinical practice, for several reasons. Fatigue-related disorders cause difficulties in memory and other cognitive function examinations. Aphasia is accompanied by cognitive deficits, which are not always easy to detect due to speech and motor impairments. Another reason is the scarcity of suitable tests that are brief yet informative. Since stroke patients are typically older, it can be assumed that memory disorders are frequent in this population. There is a bidirectional relationship between cognitive disorders and stroke. Cognitive impairment increases the risk of stroke and death, while post-stroke cognitive impairment may have existed before the stroke or may be partly caused by it. It can occur early or later after the event. Cognitive impairment persists in patients after a CVA, even after successful clinical recovery, and is closely related to poor functional outcomes.

Assessing cognitive impairment after a stroke is significant in both acute and chronic care. It helps to determine whether the patient remembers important information regarding their health status and recommendations for lifestyle changes (e.g., not smoking, adhering to a diabetic diet, regular blood pressure checks), as well as the use of essential treatments like antihypertensives or secondary preventive treatments-antiplatelet and anticoagulant therapy. Speech and memory disorders affect acute and chronic patient care-nursing, caregiving, rehabilitation, and speech therapy, as well as care in the home environment. Expressive aphasia is easily noticed, but often not quantified. Sensory aphasia is generally less recognizable from ordinary contact. The quality of the examination determines the extent of the disorder found. It is crucial for healthcare personnel to understand what to expect regarding collaboration. It is also essential to estimate whether the patient will understand the significance of the communicated information and how well they will cooperate during rehabilitation.

A physician can quickly and easily quantify speech and memory disorders after a stroke using the original Czech and innovative tests, Amnesia Light and Brief Assessment (ALBA) and Picture Naming and Immediate Recall (PICNIR). Although initially developed for patients with cognitive disorders or dementia, they are also well-suited for post-stroke patients. The validated ALBA test involves learning and repeating a six-word sentence, demonstrating six gestures according to instructions and naming them, and concluding by recalling as many words of the sentence as possible after a distraction. The validated PICNIR test consists of two parts. First, the patient names 20 black-and-white pictures. Then, the task is to recall and rewrite as many of the picture names as possible within one minute. Both tests allow for a quick and simultaneous assessment of speech and memory.

Delirium may develop in 10-30% of patients after a stroke. Post-stroke delirium may be associated with the development of cognitive impairment or dementia within three months to two years. These findings emphasize the importance of rapid detection and treatment of delirium post-stroke, as well as the monitoring of cognitive functions in subsequent years. Detecting delirium is crucial for the proper management of post-stroke care. Various tests have been developed for delirium detection. The Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) or the Intensive Care Delirium Screening Checklist (ICDSC) are commonly used. The CAM-ICU test was designed for use by both doctors and nurses in intensive care settings and has already been validated in Czech for stroke patients. While the Czech version of the ICDSC has not been validated, foreign studies suggest it is a suitable tool for delirium detection. A survey among Czech neurological departments has highlighted the need for such tests.

The investigators aim to assess the usefulness of all four methods in clinical practice for patients after a stroke. Therefore, they have prepared a project to evaluate the benefits and utilization of cognitive tests ALBA and PICNIR, and delirium tests CAM-ICU and ICDSC, in the acute phase of stroke. Additionally, they aim to validate the very short ALBA and PICNIR tests, which take less than five minutes, to improve post-stroke care in the future.

ELIGIBILITY:
Inclusion Criteria:

* Native speaker of the Czech Republic. Czech must be the patient's native language.
* Admission to the monitored bed of the neurological ICU with the possibility of initial examination within 24 hours of admission (not the onset of CVA).
* Anticipated length of hospitalization longer than five days.
* First clinical CVA in life. Subclinical signs of CVA on brain CT are acceptable.
* Absence of previous neurological deficit of any etiology affecting the brain, e.g., trauma, or spinal cord.
* Vigilant, i.e., without quantitative impairment of consciousness. Delirium may be present.

Exclusion Criteria:

* Native speaker of the Czech Republic. Czech must be the patient's mother tongue.
* Admission to the monitored bed of the neurological ICU with the possibility of initial examination within 24 hours of admission (not the onset of CVA).
* Anticipated length of hospitalization longer than five days.
* First clinical CVA in life. Subclinical signs of CVA on brain CT are acceptable.
* Absence of previous neurological deficit of any etiology affecting the brain, e.g., trauma, or spinal cord.
* Vigilant, i.e., without quantitative impairment of consciousness. Delirium may be present.
* Presence of a previous neurological deficit.
* Unfavorable prognosis upon admission.
* Discharge or anticipation of early discharge from the ICU before the follow-up examination after 5 days.
* Transient ischemic attack and conditions mimicking stroke.
* Resolution of deficit before the initial examination.
* Absence of the principal investigator.
* Intubation upon admission.
* Refusal to participate in the study by the patient or relatives.
* Complications during hospitalization affecting brain function, e.g., aspiration with hypoxia.
* Sudden progression of the condition to unconsciousness.
* Unique situations, e.g., acute endarterectomy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the monitored bed of the neurological ICU for ischemic or hemorrhagic CVA with the possibility of initial examination within 24 hours of admission (not the onset of CVA), with an anticipated length of hospitalization longer than five days, will be included in the study.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-05-03 (Estimated); Study Completion 2026-05-03 (Estimated)

PRIMARY OUTCOMES:
POBAV test | 1st day after a stroke, 5th day after a stroke
  Speech disorders after a stroke will be easily and quickly detectable using the PICNIR test, which will express the degree of impairment using numerical scales.
  In the PICNIR test, we evaluate the number of errors in pictures naming (the lower the better, preferably 0) and the number of correctly named pictures (the higher the better, max 16)
ALBA test | 1st day after a stroke, 5th day after a stroke
  Description: Speech disorders after a stroke will be easily and quickly detectable using the ALBA test, which will express the degree of impairment using numerical scales.
  ALBA score (0-12): the worst 0 and the best 12 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Fakultní Nemocnice Královské Vinohrady, Prague, Prague, Czechia

REFERENCES:
- [Background] Bartos A, Weinerova J, Diondet S. Effects of human probiotics on memory and psychological and physical measures in community-dwelling older adults with normal and mildly impaired cognition: results of a bi-center, double-blind, randomized, and placebo-controlled clinical trial (CleverAge biota). Front Aging Neurosci. 2023 Jul 7;15:1163727. doi: 10.3389/fnagi.2023.1163727. eCollection 2023. PMID 37502424
- [Background] Bartoš, A., Test ALBA byl uznán jako certifikovaná metodika Ministerstvem zdravotnictví ČR (2024) Ceska a Slovenska Neurologie a Neurochirurgie, 87 (3), p. 153.
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37502424/